CLINICAL TRIAL: NCT04785326
Title: A Randomized, Double-Blind, Multicentric, Parallel Group Therapeutic Equivalence Study Comparing Efficacy, Safety and Immunogenicity of Subcutaneous DMB-3115 and Stelara® in Patients With Moderate to Severe Chronic Plaque Psoriasis
Brief Title: Efficacy, Safety, and Immunogenicity of Subcutaneous DMB-3115 Versus Stelara® in Patients With Moderate to Severe Chronic Plaque Psoriasis
Acronym: Opportuniti
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dong-A ST Co., Ltd. (Industry)
Collaborators: Meiji Seika Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DMB-3115-2
Record Dates: First submitted 2021-03-03; First posted 2021-03-05 (Actual); Results first posted 2024-01-18 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Moderate to Severe Chronic Plaque Psoriasis
MeSH Terms: interventions — Ustekinumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- DMB-3115 (Experimental): Patients randomized to receive DMB-3115 at the beginning of the study will continue to receive the same treatment
  Interventions: Drug: DMB-3115
- Stelara (Active Comparator): Patients randomized to receive Stelara at the beginning of the study will be re-randomized at Week 28 in a 1:1 ratio to either continue on Stelara or will be transitioned to receive DMB-3115
  Interventions: Drug: DMB-3115; Drug: Stelara

INTERVENTIONS:
Drug: DMB-3115 — 45mg or 90mg dose subcutaneous administration
Drug: Stelara — 45mg or 90mg dose subcutaneous administration
  Arms: Stelara

SUMMARY:
This study is designed to evaluate efficacy, safety, pharmacokinetics (PK) and immunogenicity of subcutaneously administered DMB-3115 in comparison with Stelara for treatment of moderate to severe chronic plaque psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have a diagnosis of plaque-type psoriasis for at least 6 months.

Exclusion Criteria:

* Patients with hypersensitivity to ustekinumab or any of the product excipients.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 598 (Actual)
Dates: Start 2021-04-28 (Actual); Primary Completion 2022-02-10 (Actual); Study Completion 2022-11-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Central Sooner Research, Norman, Oklahoma
  - Jordan Valley Dermatology Center, West Jordan, Utah

RESULTS

PARTICIPANT FLOW:
Groups:
- DMB-3115: Patients randomized to receive DMB-3115 at the beginning of the study and continued to receive the same treatment
  DMB-3115: 45mg or 90mg dose subcutaneous administration
- Stelara: Patients randomized to receive Stelara at the beginning of the study and re-randomized at Week 28 in a 1:1 ratio to continue on Stelara
  Stelara: 45mg or 90mg dose subcutaneous administration
- Switch to DMB-3115: Patients randomized to receive Stelara at the beginning of the study and re-randomized at Week 28 in a 1:1 ratio to be transitioned to receive DMB-3115
  DMB-3115: 45mg or 90mg dose subcutaneous administration
  Stelara: 45mg or 90mg dose subcutaneous administration
Period: Period 1 (Week 1 to 28)
Arm/Group | DMB-3115 | Stelara | Switch to DMB-3115
Started | 299 | 299 | 0
Completed | 268 | 263 | 0
Not Completed | 31 | 36 | 0
Period: Period 2 (Week 28 to 52)
Arm/Group | DMB-3115 | Stelara | Switch to DMB-3115
Started | 268 | 132 (Period 1 Stelara Group has been re-randomized by 1:1, to Stelara group and Switch to DMB-3115 group.) | 131 (Period 1 Stelara Group has been re-randomized by 1:1, to Stelara group and Switch to DMB-3115 group.)
Completed | 258 | 130 | 124
Not Completed | 10 | 2 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DMB-3115 | Stelara | Total
Number analyzed (Participants) | 299 | 299 | 598
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.4 (13.03) | 45.7 (13.46) | 45.6 (13.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 97 | 87 | 184
  Male | 202 | 212 | 414
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Ethnicity : Hispanic or Latino | 1 | 5 | 6
  Ethnicity: Ethnicity : Not Hispanic or Latino | 297 | 294 | 591
  Ethnicity: Ethnicity : Unknown | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 3 | 0 | 3
  Race: Black or African American | 1 | 0 | 1
  Race: White | 295 | 298 | 593
  Race: Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 10 | 11 | 21
  Europe | 273 | 270 | 543
  Georgia | 3 | 2 | 5
  Ukraine | 13 | 16 | 29

OUTCOME MEASURES:

1. Primary Outcome: • To Evaluate Efficacy of DMB-3115 in Comparison With Stelara
Description: Percent change in the Psoriasis Area and Severity Index (PASI) score. PASI score is calculated by evaluating the severity of symptoms in each regions of the subject, and produces a numeric score ranging from 0 to 72.
  The higher the number, the more severe the symptoms. In general, a PASI score of 5 to 10 is considered moderate disease, and a score over 10 is considered severe.
  The primary endpoint of this clinical trial is % change in PASI, which has a value between 0 and 100, with 100 indicating complete disappearance of symptoms and 0 indicating no improvement in symptoms.
  If the patient's Baseline PASI score was 10, and 5 at the measurement period, it means that the patient showed 50% reduction.
Time Frame: Week 8 (For EMA) and 12 (For FDA)
Population: Per protocol set for EMA, Intention-to-Treat set for FDA
Measure: Least Squares Mean (Standard Error); unit: percent change in PASI score
Arm/Group | DMB-3115 | Stelara
Number analyzed (Participants) | 299 | 299
percent change in PASI score
  Week 8 (for EMA): number analyzed (Participants) | 256 | 267
  Week 8 (for EMA) | 77.5 (2.595) | 77.85 (2.587)
  Week 12 (for FDA) | 87.59 (1.886) | 87.89 (1.884)

ADVERSE EVENTS:
Time Frame: Focused primarily on treatment-emergent AEs (TEAEs), i.e., a new event that occurred during or after first dose of study treatment or any event present at baseline that worsened in either intensity or frequency after first dose of study treatment. The AEs are collected from subject's signing of informed consent until the last visit of subject, up to 57 weeks.
Description: Note that one patient of DMB-3115 group has completed period 1 and started period 2, but right after re-randomization, the subject has been withdrawn.
  So, 268 subjects of DMB-3115 group has started period 2 but the AEs are collected with 267 subjects.
Groups:
- DMB-3115 (Period 1): Patients randomized to receive DMB-3115 at the beginning of the study
  DMB-3115: 45mg or 90mg dose subcutaneous administration
- Stelara (Period 1): Patients randomized to receive Stelara at the beginning of the study
  Stelara: 45mg or 90mg dose subcutaneous administration
- DMB-3115 (Period 2): Patients randomized to receive DMB-3115 at the beginning of the study and continued to receive the same treatment
  DMB-3115: 45mg or 90mg dose subcutaneous administration
- Stelara (Period 2): Patients randomized to receive Stelara at the beginning of the study and re-randomized at Week 28 in a 1:1 ratio to continue on Stelara
  Stelara: 45mg or 90mg dose subcutaneous administration
- Switch to DMB-3115 (Period 2): Patients randomized to receive Stelara at the beginning of the study and re-randomized at Week 28 in a 1:1 ratio to be transitioned to receive DMB-3115
  DMB-3115: 45mg or 90mg dose subcutaneous administration
  Stelara: 45mg or 90mg dose subcutaneous administration
Arm/Group | DMB-3115 (Period 1) | Stelara (Period 1) | DMB-3115 (Period 2) | Stelara (Period 2) | Switch to DMB-3115 (Period 2)
All-Cause Mortality (participants affected / at risk) | 2/299 | 1/299 | 0/267 | 0/132 | 0/131
Serious Adverse Events (participants affected / at risk) | 5/299 | 3/299 | 0/267 | 2/132 | 0/131
Other Adverse Events (participants affected / at risk) | 73/299 | 90/299 | 17/267 | 15/132 | 11/131
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DMB-3115 (Period 1) (N=299) | Stelara (Period 1) (N=299) | DMB-3115 (Period 2) (N=267) | Stelara (Period 2) (N=132) | Switch to DMB-3115 (Period 2) (N=131)
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Sudden cardiac death (General disorders) | 1 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 1 | 1 | 0 | 0 | 0
COVID-19 pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Vith nerve paralysis (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DMB-3115 (Period 1) (N=299) | Stelara (Period 1) (N=299) | DMB-3115 (Period 2) (N=267) | Stelara (Period 2) (N=132) | Switch to DMB-3115 (Period 2) (N=131)
Nasopharyngitis (Infections and infestations) | 24 | 33 | 4 | 4 | 3
COVID-19 (Infections and infestations) | 14 | 18 | 4 | 2 | 3
Rhinitis (Infections and infestations) | 11 | 9 | 1 | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 4 | 11 | 3 | 1 | 0
Headache (Nervous system disorders) | 9 | 7 | 4 | 4 | 2
Hypertension (Vascular disorders) | 11 | 12 | 1 | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-06-04): https://cdn.clinicaltrials.gov/large-docs/26/NCT04785326/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-21): https://cdn.clinicaltrials.gov/large-docs/26/NCT04785326/SAP_001.pdf